CLINICAL TRIAL: NCT01513746
Title: Eating Disorders in Type 1 Diabetes: Mechanisms of Comorbidity
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00031840
Record Dates: First submitted 2012-01-17; First posted 2012-01-20 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Type 1 Diabetes; Eating Disorder
Keywords: Type 1 Diabetes; Type 1 Diabetes Mellitus; Eating Disorders; Insulin Omission
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the study is to investigate how people with type 1 diabetes experience and manage their diabetes, eating, and weight. Summary of the Study: If you choose to participate, you will complete a set of questionnaires and a structured interview. You will then wear a continuous glucose monitor and use your cell phone to answer study questions for a period of 3 days. The questions come in the form of regular phone calls between the hours of 8:00 a.m. and 10:00 p.m. Each call takes only a minute or two to complete. You will also be asked to call in and answer study questions at other times during the day, especially after eating. The study involves a minimum of 2 clinic visits to Duke. Participants who live greater than 1.5 hours from Duke can be approved to take part in the study by phone/Skype. Participants will receive and return study materials through the mail.

DETAILED DESCRIPTION:
Eating disorders (ED) are far more prevalent among individuals with type 1 diabetes (T1D) than the general population. Yet what accounts for the increased prevalence of ED in T1D, and how to effectively treat these patients is unknown. ED in T1D is dangerous. T1D patients with ED not only engage in behaviors common among non-diabetic ED patients (like binge eating), but also might omit insulin to prevent weight gain. The goal of this study is to understand the psychophysiological precipitants to ED behavior among T1D patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (aged 18-65)
2. Diagnosed with type 1 diabetes
3. Clinically significant eating disorder symptoms
4. Currently monitored by a physician

Exclusion:

1. Severe hypoglycemic unawareness
2. Pregnancy
3. Current or history of psychosis or mania
4. Current substance abuse
5. Non-English speaking
6. Significant deficits in intellectual functioning

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: UNC and Duke Endocrine Clinics Community of the Durham, Chapel Hill and Raleigh area
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2011-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Blood Glucose Values | 72 Hours

SECONDARY OUTCOMES:
Ecological Momentary Assessment of Emotional and Behavioral Outcomes | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda Merwin, PhD, Principal Investigator — Site Principal Investigator
Locations (1):
- Duke University Health System, Durham, North Carolina, United States